CLINICAL TRIAL: NCT01186328
Title: A Phase I Study Evaluating the Safety, Tolerability and Biological Activity of EZN-3042, a Survivin mRNA Antagonist, Administered With Re-induction Chemotherapy in Children With Relapsed Acute Lymphoblastic Leukemia (ALL)
Brief Title: EZN-3042 Administered With Re-induction Chemotherapy in Children With Relapsed Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enzon Pharmaceuticals decided to end its development of EZN-3042.
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2009-007
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-05

CONDITIONS: Lymphoblastic Leukemia, Acute; Lymphoblastic Leukemia, Acute, Childhood; Leukemia, Lymphoblastic, Acute, T Cell; Leukemia, Lymphoblastic, Acute
Keywords: Relapse; T cell; Lymphoblastic; Leukemia; EZN3042; Refractory; Precursor B; Pre B cell; Survivin; Acute; Childhood; Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Leukemia | interventions — EZN 3042; SPC 3042; Cytarabine; Doxorubicin; Prednisone; Vincristine; pegaspargase; Methotrexate; Hydrocortisone; hydrocortisone hemisuccinate; hydrocortisone valerate; Cortisone; hydrocortisone sodium phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will receive 2 doses of EZN-3042 (and intrathecal cytarabine, conditionally) prior to initiating systemic therapy with vincristine, doxorubicin, prednisone and PEG-asparaginase. Patients with CNS 1 or 2 will also receive intrathecal methotrexate, and patients with CNS 3 will also receive triple intrathecal therapy (methotrexate, hydrocortisone, and cytarabine).
  Interventions: Drug: EZN-3042; Drug: Cytarabine; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine; Drug: PEG-asparaginase; Drug: Methotrexate; Drug: Hydrocortisone

INTERVENTIONS:
Drug: EZN-3042 — Dose will be assigned at study entry. To be given as a 2 hour intravenous infusion on days -5, -2, 8, 15, 22 and 29. Dose levels: L0 (level zero): 1.5 mg/kg, L1: 2.5 mg/kg, L2: 5 mg/kg, L3: 6.5 mg/kg
  Other Names: SPC 3042
Drug: Cytarabine — Given intrathecally on day -6. Patients who may have received intrathecal chemotherapy within 7 days of day 0 as part of their prior maintenance chemotherapy (e.g. before the diagnosis of relapse) or as part of the diagnostic workup will not receive this dose of IT cytarabine. If given, dose is defined by age:
  1-1.99 years: 30 mg 2-2.99 years: 50 mg
  Greater than or equal to 3 years: 70 mg.
  Cytarabine is also part of the triple intrathecal therapy given to CNS 3 patients on Days 8, 15, 22 and 29. Dose is defined by age:
  1. - 1.99 years: 16 mg
  2. - 2.99 years: 20 mg
  3. - 8.99 years: 24 mg
  Greater than or equal to 9 years: 30 mg
  Other Names: ARA-C; cytosine arabinoside; Cytosar; Cytosar-U®; Arabinosylcytosine
Drug: Doxorubicin — 60 mg/m2/day given intravenous infusion (IV) over 15 minutes on day 1.
  Other Names: Adriamycin; Rubex
Drug: Prednisone — 40 mg/m2/day divided BID or TID given orally on days 1 through 29. For patients who are unable to tolerate prednisone orally, substitute IV methylprednisolone at 80% of the oral prednisone dose.
  Other Names: Prednisone Intensol®; Sterapred®; Sterapred® DS; Predone®; Deltasone®
Drug: Vincristine — 1.5 mg/m2/day (maximum dose 2 mg) given intravenous push over 1 minute or infusion via mini-bag as per institutional policy on days 1, 8, 15 and 22.
  Other Names: Oncovin®; vincristine sulfate; Vincasar Pfs®; VCR; LCR
Drug: PEG-asparaginase — 2500 IU/m2 intramuscular injection on days 2, 9, 16, 23. If available, Erwinia L-asparaginase may be substituted for pegaspargase in patients with clinically significant prior allergies to pegaspargase.
  Other Names: Oncaspar®; PEG-L-asparaginase
Drug: Methotrexate — Given intrathecally to patients with CNS1 or CNS2 disease at the dose defined by age below on days 15 and 36:
  1-1.99 years: 8 mg 2-2.99 years: 10 mg 3-8.99 years: 12 mg
  Greater than or equal to 9 years: 15 mg
  Given as part of the Triple intrathecal therapy to patients with CNS 3 disease at the doses defined by age below on days 8, 15, 22 and 29:
  1. - 1.99 years: 8 mg
  2. - 2.99 years: 10 mg
  3. - 8.99 years: 12 mg
  Greater than or equal to 9 years: 15 mg
  Other Names: Rheumatrex; Trexall; Amethopterin; Methotrexate Sodium; MTX
Drug: Hydrocortisone — Given as part of the Triple intrathecal therapy to patients with CNS 3 disease at the doses defined by age below on days 8, 15, 22 and 29:
  1. - 1.99 years: 8 mg
  2. - 2.99 years: 10 mg
  3. - 8.99 years: 12 mg
  Greater than or equal to 9 years: 15 mg
  Other Names: Ala-Cort ®; Hydrocortone Phosphate; Solu-Cortef®; Hydrocort Acetate®; Lanacort®; Cortef®; Westcort®; Cortisone; Hydrocortisone Sodium Succinate; Hydrocortisone Sodium Phosphate

SUMMARY:
An experimental drug called EZN-3042 targets survivin, a protein expressed in leukemia cells at relapse that promotes the leukemia cells to grow. The main goal of this phase I study is to find out the dose of EZN-3042 that can be safely given without serious side effects both alone and in combination with standard chemotherapy drugs during re-induction.

DETAILED DESCRIPTION:
This is a phase I multi-site study of the new investigational agent EZN-3042, which is highly effective at blocking survivin and inhibiting survivin protein expression. Survivin plays pivotal roles in tumor formation by inhibiting cell death and regulating cell cycle progression. The primary objective is to study EZN-3042 in children with relapsed acute lymphoblastic leukemia (ALL). Patients will receive 2 doses of EZN-3042 (and intrathecal cytarabine, conditionally) prior to initiating systemic therapy with vincristine, doxorubicin, prednisone and PEG-asparaginase. Patients with CNS 1 or 2 will also receive intrathecal methotrexate, and patients with CNS 3 will also receive triple intrathecal therapy (methotrexate, hydrocortisone, and cytarabine). Blood and bone marrow specimens will be drawn to measure minimal residual disease (MRD), pharmacokinetic levels of EZN-3042 and survivin expression. The study will follow a standard 3+3 dose escalation design. We hypothesize that EZN-3042 will be safe, tolerable and biologically active, when given both alone and in combination with standard re-induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥1 and ≤ 21 years of age when originally diagnosed with acute lymphoblastic leukemia (ALL).
* Patients must have relapsed or refractory B-precursor acute lymphoblastic leukemia (ALL) with ≥25% blasts in the bone marrow (M3), with or without extramedullary disease.
* Patients may have central nervous system 1, 2 or 3 disease.
* Karnofsky Performance Level ≥ 50 for patients > 10 years of age and Lansky ≥ 50 for patients ≤ 10 years of age.
* Patients must have had 2 or more prior therapeutic attempts defined as:

  * Relapse after going into remission from re-induction for the first or subsequent relapse (ie: 2nd , 3rd, 4th…relapse), or
  * Refractory disease after first or greater relapse and a single re-induction attempt. *Please note, Enrollment will be restricted to at most one refractory patient in each cohort of 3 patients per dose level.
  * Patients with ALL who are refractory to frontline induction therapy are not eligible.
* Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study.
* Patients who relapse when they are not receiving standard ALL maintenance therapy must have fully recovered from grade 3 or 4 toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Cytotoxic Therapy: It must be at least 14 days since the completion of cytotoxic therapy (excluding hydroxyurea) at the time of study enrollment.
* Hematopoietic Stem Cell Transplant (HSCT): Patients who have experienced their relapse after a HSCT are eligible, provided they have no evidence of active Graft-versus-Host Disease (GVHD) and are at least 120 days post-transplant at the time of enrollment.
* Prior anthracycline exposure: Patients must have ≤ 400 mg/m2 lifetime exposure of anthracycline chemotherapy.
* Biologic (anti-neoplastic) therapy: It must be at least 7 days since the completion of therapy with a biologic agent at the time of study enrollment. For agents that have known adverse events occurring 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
* Patients must have a calculated creatinine clearance or radioisotope GRF ≥ 70mL/min/1.73m2 OR a normal serum creatinine based on the institutional normal values according to age.
* Patient's ALT must be < 5 x institutional upper limit of norm (ULN), unless the elevation is suspected to be disease-related.
* Patient's total bilirubin must be ≤ 1.5 x ULN.
* Patient's serum albumin must be ≥ 2 g/dL.
* Patient must have prothrombin time (PT), partial thromboplastin time (PTT) and international normalized ratio (INR) ≤ 1.5 times the ULN.
* Patient must have a shortening fraction ≥ 27% by echocardiogram or an ejection fraction ≥ 45% by gated nucleotide study.
* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

Exclusion Criteria:

* Patients with Down syndrome are excluded.
* Patients with B-cell ALL (L3 morphology or evidence of myc translocation by molecular or cytogenetic technique) are not eligible
* Patients who cannot receive asparaginase on this study due to prior pancreatitis, stroke or other toxicity are not eligible.

  * Patients with clinically significant prior allergies to PEG asparaginase are eligible if Erwinia L-asparaginase can be substituted. The study will not supply Erwinia.
  * Patients who initially receive asparaginase, but must discontinue due to toxicity, remain eligible.
* Patients with documented active and uncontrolled infection at the time of study entry are not eligible.
* Patient will be excluded if they are currently receiving other investigational drugs.
* Patients will be excluded if they are taking strong CYP3A4 inducers or inhibitors.
* Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2010-08-24 (Actual); Primary Completion 2012-01-10 (Actual); Study Completion 2012-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raetz, MD, Study Chair — NYU Langone Health; William Carroll, MD, Study Chair — NYU Langone Health
Locations (7):
- United States (6):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - New York University Medical Center, New York, New York
  - St. Jude, Memphis, Tennessee
- Sydney Children's Hospital, Sydney, Australia

REFERENCES:
- [Result] Raetz EA, Morrison D, Romanos-Sirakis E, Gaynon P, Sposto R, Bhojwani D, Bostrom BC, Brown P, Eckroth E, Cassar J, Malvar J, Buchbinder A, Carroll WL. A phase I study of EZN-3042, a novel survivin messenger ribonucleic acid (mRNA) antagonist, administered in combination with chemotherapy in children with relapsed acute lymphoblastic leukemia (ALL): a report from the therapeutic advances in childhood leukemia and lymphoma (TACL) consortium. J Pediatr Hematol Oncol. 2014 Aug;36(6):458-63. doi: 10.1097/MPH.0b013e3182a8f58f. PMID 24276047
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients were initially enrolled onto Dose Level 1. 1 of 3 patients were found to experience a dose limiting toxicity. 3 additional patients were enrolled onto dose level 1. Another 1 patient was found to experience a DLT that was deemed possibly related to study medication EZN-3042. Study dose was deescalated to dose level 0.
Groups:
- EZN Dose Level 1: Dose Level 1 is the starting dose level. Patients will receive 2 doses of EZN-3042 at 2.5 mg/m2/day (and intrathecal cytarabine, conditionally) prior to initiating systemic therapy with vincristine, doxorubicin, prednisone and PEG-asparaginase, and then Day 8, 15, 22, and 29. If MTD is exceeded at dose level 1, the dose level will be deescalated to Dose Level 0.
- EZN Dose Level 2: If the MTD is not exceeded at dose level 1, the dose will be escalated to dose level 2 at 5mg/m2/day. Dose will be administered following the same dosing schedule as Dose level 1.
- EZN Dose Level 3: If the MTD is not exceeded at Dose Level 2, the dose will be escalated to Dose Level 3 at 6.5 mg/kg following the same dosing schedule as Dose Level 1 and 2.
Period: Overall Study
Arm/Group | EZN Dose Level 1 | EZN Dose Level 2 | EZN Dose Level 3
Started | 6 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | EZN Dose Level 1
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Prior HSCT [Count of Participants; unit: Participants]
  Yes | 2
  No | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of EZN-3042
Description: To determine the recommended dose of EZN-3042 administered weekly in combination with re-induction chemotherapy. Based on disease response at Day 36 and toxicity profile assessed until 30 days after discontinuation of study drug.
Time Frame: 2 months
Population: 6 patients were enrolled at Dose Level 1. Dose level deescalated to Dose level 0 after 2 patients in Dose Level 1 experienced dose limiting toxicities. No patients were accrued on Dose level 0 prior to study closure.
Measure: Count of Participants; unit: Participants
Groups:
- EZN Dose Level 0: Study deescalated to Dose Level 0 at 1.5 mg/kg after 2 patients at Dose Level 1 experienced DLTs.
Arm/Group | EZN Dose Level 1 | EZN Dose Level 0
Number analyzed (Participants) | 6 | 0
Participants
  Completed therapy w/o DLT | 4 | 0
  Experienced DLT | 2 | 0

2. Secondary Outcome: Number of Participants Who Showed a Decrease From Day -6 in Survivin Transcript Expression After EZN-3042 Administration
Description: To evaluate primary target engagement of EZN-3042 we will examine survivin transcript and protein expression before (Day -6) and after EZN-3042 administration (Day 0) in enriched bone marrow blasts in children with relapsed B-precursor leukemia.
Time Frame: Day -6 to Day 0
Population: Five patients provided samples for pharmacokinetic analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | EZN Dose Level 1
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: 11 months
Description: The definitions of AE and SAE used to collect information do not differ from the clinicaltrials.gov definitions.
Arm/Group | EZN Dose Level 1
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EZN Dose Level 1 (N=6)
Aspartate aminotransferase increased (Investigations) | 1
GGT increased (Investigations) | 1
Lung infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EZN Dose Level 1 (N=6)
Abdominal pain (Gastrointestinal disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Patient presented with pancreatitis, u/s revealed colonic pneumatosis.
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 — ferritin=11,000ug/ml on 05/17/11. Hemosiderosis per liver biopsy
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infusion site extravasation (General disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Blood and lymphatic system disorders) | 4
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Serum amylase increased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Metabolism and nutrition disorders) | 4
White blood cell decreased (Blood and lymphatic system disorders) | 5

LIMITATIONS AND CAVEATS:
The study was terminated early because Enzon Pharmaceuticals decided to halt development of EZN-3042.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days